CLINICAL TRIAL: NCT05458752
Title: Pneumocystis Jirovecii Pneumonia in Non-HIV-infected Immunocompromised Patients : a Prognostic Observational Retrospective Monocentre Study
Brief Title: Pneumocystis Jirovecii Pneumonia in Non-HIV-infected Immunocompromised Patients
Acronym: PnP-HIV-Free
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, LEFEVRE Benjamin, Doctor, Central Hospital, Nancy, France
Other Study IDs: 2020PI184-Pre-existing datas
Record Dates: First submitted 2022-06-28; First posted 2022-07-14 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-07

CONDITIONS: Pneumocystis Jirovecii Infection
Keywords: pneumocystis jirovecii pneumonia; HIV-free patients
MeSH Terms: conditions — Pneumocystis Infections; Pneumonia, Pneumocystis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Pneumocystis jirovecii pneumonia (PjP) is a rare infectiouse disease with a high level of mortality. PjP is a classical opportunistic infection which concern HIV infected and immunocompromised patients. During the past decade, several therapeutic's progresses have been done in oncology, immunology and hematology. As a consequence, patients benefited of greater treatment efficacy but are exposed to a higher risk of opportunistic infections as PjP. The investigators hypothesis is that PjP incidence increase and its form is depending of underlying immune conditions. The investigators aim to describe its incidence, the PjP forms depending on comorbidities and to identifiy pronostics factors.

ELIGIBILITY:
Inclusion Criteria:

* Underlying immune condition at risk of Pneumocystis jirovecii pneumonia excluding HIV infection
* Clinical, biological and radiological presentation which evoke Pneumocystis jirovecii pneumonia
* Microbiological confirmation by respiratory specimen analyses ( specific coloration and/or IFI and/or PRC)

Exclusion Criteria:

* No microbiological confirmation by respiratory specimen analyses
* Proved HIV infection
* Patient denied to particpate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients without HIV-infection hospitalised in Nancy hospital between 2004 and 2021 for Pneumocystis jirovecii pneumonia
Sampling Method: Non-Probability Sample
Enrollment: 133 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Incidence of Pneumocystis jirovecii pneumonia in HIV-free patients | Between the first january 2004 and the 31th december 2021
  Number of cases / number of patients treated for a predisposing disease (heamotological or imunological disease, or cancer...)

SECONDARY OUTCOMES:
To describe the age of giv free patients with Pneumocystis jirovecci pneumonia | Between the first january 2004 and the 31th december 2021
  age in years
To describe the body mass index of HIV free patients with Pneumocystis jirovecci pneumonia | Between the first january 2004 and the 31th december 2021
  BMI in kg/m2 (quanti
To describe the Charlson comorbidity index of HIV free patients with Pneumocystis jirovecci pneumonia | Between the first january 2004 and the 31th december 2021
  Charlson comorbidity index as a quantitative variable
To describe the comoribidites of HIV-free patients with Pneumocystis jirovecci pneumonia | Between the first january 2004 and the 31th december 2021
  Comorbidities as categorial variables
To describe the previous medications used by HIV free patients with Pneumocystis jirovecci pneumonia | Between the first january 2004 and the 31th december 2021
  Medications as categorial variables
To describe clinical features of Pneumocystis jirovecci pneumonia in HIV-free patients | Between the first january 2004 and the 31th december 2021
  Type of first symptoms as categorial variables
To describe the date of the first symptoms of Pneumocystis jirovecci pneumonia in HIV-free patients | Between the first january 2004 and the 31th december 2021
  Date of first symptoms as quantitative variable
To describe the pO2 level of HIV free patients with Pneumocystis jirovecci pneumonia | Between the first january 2004 and the 31th december 2021
  pO2 (in mmHg)
To describe the PCR level of HIV free patients with Pneumocystis jirovecci pneumonia | Between the first january 2004 and the 31th december 2021
  PCR (mg/L)
To describe the WBC level of HIV free patients with Pneumocystis jirovecci pneumonia | Between the first january 2004 and the 31th december 2021
  WBC (G/L)
To describe the creatinine level of HIV free patients with Pneumocystis jirovecci pneumonia | Between the first january 2004 and the 31th december 2021
  Creatinine (µmol/L)
To describe the LDH level of HIV free patients with Pneumocystis jirovecci pneumonia | Between the first january 2004 and the 31th december 2021
  LDH (MUI/L)
To describe the albumin level of HIV free patients with Pneumocystis jirovecci pneumonia | Between the first january 2004 and the 31th december 2021
  albumin (g/L)
To describe the immunoglobulin level of HIV free patients with Pneumocystis jirovecci pneumonia | Between the first january 2004 and the 31th december 2021
  immunoglobulin (g/L)
To describe the lymphocytes level of HIV free patients with Pneumocystis jirovecci pneumonia | Between the first january 2004 and the 31th december 2021
  lymphocytes (G/L)
To describe the PCR pneumocystis level of HIV free patients with Pneumocystis jirovecci pneumonia | Between the first january 2004 and the 31th december 2021
  PCR pneumocystis in ct
To describe the immunofluorescence value of HIV free patients with Pneumocystis jirovecci pneumonia | Between the first january 2004 and the 31th december 2021
  Immunofluorescence as a categorial variable
To describe the specific coloration value of HIV free patients with Pneumocystis jirovecci pneumonia | Between the first january 2004 and the 31th december 2021
  Specific coloration as a categorial variable
To describe the use of nasal canula in HIV free patient with a Pneumocystis jirovecci pneumonia | Between the first january 2004 and the 31th december 2021
  Nasal canula as a categorial variable
To describe the use of high flow oxygenation in HIV free patient with a Pneumocystis jirovecci pneumonia | Between the first january 2004 and the 31th december 2021
  High flow oxygenation as a categorial variable
To describe the use of mechanical ventilation in HIV free patient with a Pneumocystis jirovecci pneumonia | Between the first january 2004 and the 31th december 2021
  Mechanical ventilation as a categorial variable
To describe the duration of hospitalisation of HIV free patients with Pneumocystis carinii pneumonia | Between the first january 2004 and the 31th december 2021
  Duration in days
To describe the use of cotrimoxazole for HIV free patients with Pneumocystis carinii pneumonia | Between the first january 2004 and the 31th december 2021
  cotrimoxazole as a categorial variable
To describe the use of atovaquone for HIV free patients with Pneumocystis carinii pneumonia | Between the first january 2004 and the 31th december 2021
  atovaquone as a categorial variable
To describe the use of pentamidine for HIV free patients with Pneumocystis carinii pneumonia | Between the first january 2004 and the 31th december 2021
  pentamidine as a categorial variable
To describe the use of steroïd for HIV free patients with Pneumocystis carinii pneumonia | Between the first january 2004 and the 31th december 2021
  steroïd as a categorial variable

CONTACTS AND LOCATIONS:
Locations (1):
- Université de Lorraine, CHRU Nancy and APEMAC, Vandœuvre-lès-Nancy, Lorraine, France

IPD SHARING:
Plan to Share IPD: No